CLINICAL TRIAL: NCT03710720
Title: Mentorship and Research in HIV and Addiction Prevention Among Traumatized Youth
Brief Title: Trauma Informed Prevention for Substance Use and Risky Sex
Acronym: TIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00041527
Record Dates: First submitted 2018-10-15; First posted 2018-10-18 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Substance Use; HIV/AIDS
Keywords: Traumatic stress; substance use prevention; HIV prevention; adolescents
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Urn randomization will be monitored by the Principal Investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TF-CBT plus TIPS app (Experimental)
  Interventions: Behavioral: TIPS app; Behavioral: Trauma Focused-Cognitive Behavioral Therapy
- TF-CBT (Active Comparator)
  Interventions: Behavioral: Trauma Focused-Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: TIPS app — Psycho-educational electronic application
  Arms: TF-CBT plus TIPS app
Behavioral: Trauma Focused-Cognitive Behavioral Therapy — Effective form of trauma therapy for adolescents
  Other Names: TF-CBT

SUMMARY:
The purpose of this research study is to determine the usefulness of the TIPS iPad app in the treatment of adolescent patients who qualify for Trauma Focused-Cognitive Behavioral Therapy (TF-CBT).

DETAILED DESCRIPTION:
The primary goal of this study is to conduct a feasibility test of the delivery of the TIPS app during implementation of TF-CBT in comparison to TF-CBT as it is usually administered, as well as feasibility of methods that would be utilized in a larger scale evaluation of the toolkit. Clients will be randomly assigned to one of the two conditions, TF-CBT plus the TIPS app or TF-CBT as usual. Study duration is six months and includes four total assessments, which will be completed by hand. These assessments will occur over the 12-16 weeks of TF-CBT that clients would receive whether they choose to participate in the study or not. Participation in this study may broaden your child's treatment to target prevention of risk behaviors, but that cannot be guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* Have experienced at least one traumatic event

Exclusion Criteria:

* Adolescents exhibiting psychotic symptoms
* Significant cognitive disability
* PDD
* Active suicidal or homicidal ideations
* Meets criteria for a DSM-5 moderate or severe substance use disorder

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Risky Sexual Behaviors Scale | Pretreatment to 6 month follow-up
  The Risky Sexual Behaviors Scale (RSBS) is a validated measure that was originally created to gain more insight on the behaviors of a population of homeless adolescents. The scale measures increased risk of STDs through four major scale items. The RSBS uses a five-point Likert scale that targets caregiver involvement in discussions surrounding sexual behaviors with the option for least involved being "never" (score of 1) and the greatest involved being "always" (score of 5). The scale also includes fill-in-the-blank questions that gauge the number of "times" an adolescent has engaged in a specific behavior in the past 30 days and the past 90 days. Higher scores are indicative of higher rates of risky sexual behaviors.

SECONDARY OUTCOMES:
Family Environment Scale | Pretreatment to 6 month follow-up
  The Family Environment Scale (FES) is a validated measure that is made up of 26 "true or false" questions that target different interactions that commonly occur within families. We are using two validated subscales from this measure, family conflict and family cohesion. Higher scores on the family conflict subscale are indicative of greater rates of family conflict. Higher rates on the family cohesion subscale are indicative of higher rates of family cohesion. The measure aims to detect an increase in positive family environment over time.
Bad Friends Subscale of the Pittsburgh Youth Study | Pretreatment to 6 month follow-up
  The Bad Friends Subscale of the Pittsburg Youth Study (Youth-Friends Scale) is a validated measure made up of eight questions (both fill-in-the-blank and yes/no) that aim to detect caregiver approval of adolescent peer groups and whether caregiver opinions are considered in future peer interactions. The scale aims to detect a decrease in negative peers over time. Answers are qualitative in nature. In general, the rater looks for themes in regards to whether the youth spends time with negative peers (that the caregiver does not approve of).
Alabama Parenting Questionnaire | Pretreatment to 6 month follow-up
  The Alabama Parenting Questionnaire (APQ) is a validated measure consisting of questions that look into family interactions and, more specifically, interactions between youth and caregiver. The scale is scored on a five-point Likert scale that ranges from "never" (score of 1) to "always" (score of 5) when looking at how often certain behaviors occur within the home. High scores on the positive parenting subscale and low scores on the poor monitoring/supervision, inconsistent discipline, and corporal punishment subscales are indicative of positive parenting.
UCLA PTSD Index DSM-V | Pretreatment to 6 month follow-up
  The UCLA Post Traumatic Stress Disorder Index DSM-IV (UCLA PTSD Index DSM-IV) is a validated, subjective measure that consists of 23 yes or no questions regarding the occurrence of different traumas or losses that may happen during a child's life. Each question is followed up with details of the trauma that occurred and more extensive questioning for the trauma experienced that is still most bothersome in the present day. These follow-up questions gauge symptoms of PTSD on a five-point Likert scale that ranges from "none" (score of 0, no days has this symptom occurred in the last month) to "most" (score of 4, symptom occurred almost every day in the past month). The most traumatic experience is also followed by several yes/no questions that gauge distress and functional impairment. Higher scores are indicative of higher rates of PTSD symptoms.
Children's Depression Inventory | Pretreatment to 6 month follow-up
  The Children's Depression Inventory (CDI) is a validated measure that consists of 27 multiple choice items that gauge depressive behaviors/symptoms in youth. The items each have three choices that are best described as "Never/Rarely," "Many," or "All" in regards to each behavior in question. Higher scores are indicative of higher rates of depressive symptoms.
Timeline Follow Back (TLFM)-Form 90 | Pretreatment to 6 month follow-up
  The Timeline Follow Back (TLFB) is a validated, subjective measure that uses a calendar for people to provide estimates of substance use (drugs/alcohol) on a daily basis, retrospectively. Key dates and calendars are used to aid in memory recall. The measure is beneficial in both clinical and research environments. Over time, the TLFB looks for a decrease in alcohol use. Higher numbers of substance use are indicative of greater substance use.
CRAFFT Screening Tool for Adolescent Substance Abuse | Pretreatment to 6 month follow-up
  Scores of two or more are indicative of a probable substance use problem.

CONTACTS AND LOCATIONS:
Overall Officials: Carla K Danielson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Danielson CK, Moreland A, Hahn A, Banks D, Ruggiero KJ. Development and Usability Testing of an mHealth Tool for Trauma-Informed Prevention of Substance Use, HIV Acquisition, and Risky Sexual Behaviors Among Adolescents: Mixed Methods Study. JMIR Form Res. 2024 Jan 18;8:e52835. doi: 10.2196/52835. PMID 38236634